CLINICAL TRIAL: NCT06039332
Title: Subjective and Audiological Benefit of BONEBRIDGE (BCI602) With Two Different Fitting Strategies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario La Paz (Other)
Collaborators: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Principal Investigator, Miryam Calvino, Investigator, Member of the Research Department, Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI-6471
Record Dates: First submitted 2023-08-25; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Bone Conduction Deafness; Quality of Life; Hearing Loss, Mixed
MeSH Terms: conditions — Hearing Loss, Mixed Conductive-Sensorineural

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fittig with DSL-BCD (Experimental): The new way of fitting the audioprocessor
  Interventions: Procedure: Fitting of the audioprocessor with the auditory implant BCI602
- Fitting with DSL v5 (Active Comparator): The way of fitting the audioprocessor until now
  Interventions: Procedure: Fitting of the audioprocessor with the auditory implant BCI602

INTERVENTIONS:
Procedure: Fitting of the audioprocessor with the auditory implant BCI602 — to compare the performance with BB system in two fitting-configurations (active comparator: DSL v5, experimental: DSL-BCD) using audiometric and subjective measures

SUMMARY:
The Bonebridge (BB) is a partially implantable active transcutaneous bone conduction hearing system manufactured by MED-EL Elektromedizinische Geräte Gesellschaft m.b.H. (MED-EL, Innsbruck, Austria).

The BB augments hearing by providing acoustic input to the inner ear via bone conduction.

In 2017 Hodgetts & Scollie introduced a new fitting algorithm called DSL-BCD. The DSL-BCD algorithm was developed especially for the characteristics of bone conduction devices (BCD). If there is a benefit on the patient level in hearing outcomes when comparing the application of DSL-BCD in comparison to DSL v5 when using the BB, was not yet investigated.

The aim of this clinical study is to show the improvement in audiological performance and subjective satisfaction with the BCI602 and SAMBA 2 audio processor in patients with conductive hearing loss compared to the unaided condition and to evaluate performance differences through application of 2 different fitting algorithms, namely DSL v5 and DSL-BCD.

DETAILED DESCRIPTION:
1. The objective of this study was to verify the influence of different fitting procedures
2. Duration of investigation:

   Unexperienced users group: Each subject will be actively involved in the study for a period of 4-6 weeks after the first fitting of the audio-processor, 4 visits in total.

   Experienced users group: Each subject implanted for at least 3 months will be asked to be involved in the study the day of their following scheduled fitting, 1 visit in total.

   We expect the study to conclude within 3 years for study start.
3. Study design: The study is designed as a prospective two-period crossover, single-subject repeated-measures. It is intended to compare the performance with and without BB system in two fitting-configurations (A: DSL v5, B: DSL-BCD) using audiometric and subjective measures. For evaluation each subject serves as his/her own control. For experienced users only acute tests in condition A and B (order randomised, sequence AB or BA) will take place. For unexperienced users the period with each condition will be 2 to 3 weeks. From the clinical perspective no specific washout period between fitting A and B is needed to avoid a carryover effect. Heterogeneity and variability inherent to the population and their outcome measures will be recognized. By using a single-subject design, the effect of variability is minimized. The use of standardized evaluation methods assures the reliability of the data across investigational center.
4. Randomisation: To eliminate the sequence effect, we performed a block randomisation to ensure that the number of patients in each sequence (fitting with configuration A or B) is similar throughout the study.
5. Inclusion criteria:

   * 18 years of age or older
   * Unilateral and/or bilateral CHL/MHL in the device indication range
   * Implanted with a BCI602 device
   * Willingness and ability to use the hearing system and to perform all tests required for the study
   * Signed, and dated informed consent before the start of any study specific procedure
   * Native speaker 5.1. Exclusion criteria: A patient with/is
   * Profound unilateral sensorineural hearing loss, often termed Single Sided deafness (SSD)
   * retrocochlear, or central auditory disorders
   * any physical, psychological, or emotional disorder that would interfere with the ability to perform on test and rehabilitation procedures
   * fluctuating hearing loss
   * subjects who do not meet one or more of the above mentioned inclusion criteria are excluded from the study
6. Fitting:

Fitting condition A: Fitted on study audioprocessor: DSL v5, Acclimatization Level - 100%, First Fit Fitting condition B: Fitted on study audioprocessor: simulated DSL-BCD, simulated on the basis of DSLv5 with adjustments to reach the DSL-BCD Only used in the experienced user group: Fitting condition C: Patients own fitting, with adjustments for best fit, fitted on patients own audioprocessor

7. Study procedure:

Test intervals Prospective design: Subjects will be evaluated in four intervals.

1. st Session The first session takes place before surgery.
2. nd Session The 2nd session will take place at activation of the Bonebridge hearing system.
3. rd Session The 3rd session will take place after 2-3 weeks using the Bonebridge in the first fitting condition.
4. th Session The 4th session will take place after 2-3 weeks using the Bonebridge in the second fitting condition.

Retrospective design: Subjects will be evaluated in one interval.

1. st Session The only session takes place the day of the next scheduled fitting (at least 3 months later their first fitting). Patient will be evaluated with their current fitting (DSL v5), and the new fitting condition (DSL-BCD).

   The 1st session comprises the following tests:

   o unaided: Speech and Spatial Questionnaire (SSQ12) / Abbreviated Profile of Hearing Aid Benefit (APHAB)

   o Air conduction/Bone conduction under headphone, bilaterally

   o Sound field tone audiometry with warble tone in unaided condition
   * Sound field speech in quiet testin unaided condition
   * Sound field speech in noise in unaided condition

   The 2nd session (acute measurements) comprises the following tests:

   o BC threshold measurement, bilaterally

   o Sound field tone audiometry with warble tone in aided condition, condition A & B*

   o Sound field speech in quiet test in aided condition, condition A & B*

   o Sound field speech in noise in aided condition, condition A & B*

   o Preference A or B questionnaire

   o SAMBA 2 will be handed out with the fitting condition according to the randomization plan * If the randomization plan provides the patient with fitting condition B for the first 2-3 weeks, then condition B will be measured first in all acute sound field measurements at visit 2.

   The 3rd session (after 2-3 weeks of use) comprises the following tests:

   o Optional: BC threshold measurement, bilaterally

   o Aided: questionnaires SSQ12 / APHAB

   o Wearing time will be noted
   * Sound field tone audiometry with warble tone in aided condition , unaided & condition A*
   * Sound field speech in quiet test in aided condition, unaided & condition A*
   * Sound field speech in noise in aided condition, unaided & condition A*
   * SAMBA 2 will be handed out with the fitting condition according to the randomization plan

   The 4th session (after another 2-3 weeks of use) comprises the following tests:

   o Aided: questionnaires SSQ12 / APHAB
   * Wearing time will be noted
   * Sound field tone audiometry with warble tone in aided condition, condition B* & acute in condition A
   * Sound field speech in quiet test in aided condition, condition B* & acute in condition A
   * Sound field speech in noise in aided condition, condition B* & acute in condition A
   * Preference A or B questionnaire
   * Release of the patient from the study followed by personalized fitting of BB for the patient

     8. Data Management: The data manager will have the following duties and assure: Data anonymity, data management and reporting of data capture, follow conclusions set out in the study protocol and can be reliably drawn from the database. Concerns are identified and reported accurately. Creates a database, validates a database, documents data received. Performs database entry and processing, validation of entered data, data entry errors, and operates database security.

   Available data from patients who dropped out of the study at a certain time point or who are lost to follow-up will be used for analysis. Source data will be verified by the investigator.

   Data of participants will be pseudonymised for data handling and analysis and anonymised for publication.

9. Statistical Analysis Descriptive statistics: To be used to report demographic (e.g. age and gender) and baseline characteristics (e.g. aetiologies). Quantitative data will be presented as mean, standard deviation and range (minimum and maximum); qualitative data as in questionnaires will be presented as absolute and relative frequencies and if appropriate as graphs. Parametric Student's t-tests or nonparametric Wilcoxon signed rank tests will be performed, depending on the data distribution. Kolmogorov-Smirnov test will be used to check for data distribution.Two-period crossover data analysis: General Linear Models with "time" (visit 3 vs. visit 4) and "treatment" (fitting A vs. fitting B) as fixed factors will be used to analyze the time-by-treatment interaction for each tested hearing outcomes. Additionally, to verify the assumption that there is no sequence effect, the mean of the dependent variables (e.g. speech test outcomes, sound field thresholds) will be compared between the AB (difference between B and A) and BA (difference between A and B) sequences.

Handling of missing data: Missing data will not be replaced but treated as "missing" values. Statistical significance will be set to p<0.05. SPSS software will be used for all analyses. Graphs will be created in Microsoft Office Excel.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Unilateral and/or bilateral conductive or mixed hearing loss (CHL/MHL) in indication range.
* Implanted with a BCI602 device.
* Willingness and ability to use the hearing system and to perform all tests required for the study
* Signed, and dated informed consent before the start of any study specific procedure
* Native speaker

Exclusion Criteria:

* Profound unilateral sensorineural hearing loss, often termed Single sided deafness (SSD)
* Retrocochlear, or central auditory disorders
* Any physical, psychological, or emotional disorder that would interfere with the ability to perform on test and rehabilitation procedures
* Subjects who do not meet one or more of the above mentioned inclusion criteria are excluded from the study.
* Fluctuating hearing loss.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-27 (Estimated)

PRIMARY OUTCOMES:
Audiological performance with both ways of fitting | 12 weeks
  Standard audiometry Sound field testing will be conducted in quiet with the subject sitting one meter from the loudspeakers. The volume control of the device shall be set at the most comfortable level for the sound field tests.
Speech performance in quiet with both ways of fitting | 12 weeks
  Speech audiometry in quiet The word recognition score will be measured in quiet. The test in quiet shall be conducted with the speaker at 0° azimuth (S0) with 1 meter distance from the center of the subject's head and at ear level.
  Spanish speech material (recorded): Cardenas and Marrero balanced word list. 100% will be considered as the maximum outcome
Speech performance in noise with both ways of fitting | 12 weeks
  Speech audiometry in noise For measuring speech intelligibility in noise the International Matrix Test is used with fixed noise level at 65 dB SPL and speech level at 65 dB SPL from S0N0 (speech and noise coming from the front). One list comprises 20 sentences with 5 words in each sentence. A negative value means, better performance
Subjective satisfaction measured with SSQ12 | 12 weeks
  Questionnaires
  A hearing specific questionnaire will be filled out per participant, in 3 conditions, unaided (preoperatively), aided with BB in fitting condition A and aided with Bonebridge in fitting condition B.
  The Spanish version of Speech, Spatial, and Qualities of Hearing Questionnaire with 12 items (SSQ12) will be used. It is designed to measure self-reported auditory disability across a wide variety of domains, reflecting the reality of hearing in the everyday world. It takes approximately 5 minutes to complete. It consists of 12 questions that the subjects score on a scale from 0 (not at all) to 10 (perfectly). The total score is the sum of all items and can range between 0 and 120. The higher score, the better outcomes.
Subjective satisfaction evaluated by means of APHAB | 12 weeks
  Questionnaires A hearing specific questionnaire will be filled out per participant, in 3 conditions, unaided (preoperatively), aided with BB in fitting condition A and aided with Bonebridge in fitting condition B.
  The Spanish version the Abbreviated Profile of Hearing Aid Benefit (APHAB) will be used.
  It is a 24-item questionnaire derived from the original 66-item Profile of Hearing Aid Benefit. The self-assessment instrument evaluates hearing impairment in real-life situations with and without hearing aids. Participants have to rate how often a given statement is true in their daily life, based on the following seven response alternatives: always (99%), almost always (87%), generally (75%), half-the-time (50%), occasionally (25%), seldom (12%) and never (1%). In the first three subscales, higher scores suggest less hearing disability, while lower scores indicate less hearing disability in the aversiveness subscale. The APHAB typically requires 10 minutes or less to complete.
Subjective satisfaction assessed by a custom made questionnaire | 12 weeks
  Questionnaires A hearing specific questionnaire will be filled out per participant, in 3 conditions, unaided (preoperatively), aided with BB in fitting condition A and aided with Bonebridge in fitting condition B.
  A third, custom made questionnaire, will be filled out at two timepoints, after the acute test of condition A & B in visit 2 and at the last visit. The questionnaire will ask the patient what condition A or B was preferred in visit 2. At the last visit (for the unexperienced users, and in the only visit for the experienced users) the patient will be asked what condition was preferred in several listening scenarios during the trial time.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Gavilan, Study Chair — Hospital La Paz
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No